CLINICAL TRIAL: NCT03152864
Title: Stabilizing Behavioral Rhythms to Improve Mental Health
Acronym: SRMH
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: HealthRhythms, Inc. (Industry)
Collaborators: National Institute of Mental Health (NIMH) (NIH); University of Utah (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1R44MH113520 (NIH); R44MH113520 (NIH)
Record Dates: First submitted 2017-04-24; First posted 2017-05-15 (Actual); Last update posted 2021-07-01 (Actual); Status verified 2021-06

CONDITIONS: Depressive Symptoms; Anxiety Symptoms; Sleep Symptoms
MeSH Terms: conditions — Depression; Anxiety Disorders

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Full Package (Experimental)
  Interventions: Behavioral: Full Package
- Sensing Only (No Intervention)

INTERVENTIONS:
Behavioral: Full Package — Individuals will be randomly allocated to receive the full HealthRhythms package (Rhythm Sensing, Rhythm Trending, and Rhythm Stabilization) program on their smartphones
  Arms: Full Package

SUMMARY:
In order to assess the efficacy of the Rhythm Stabilization component of HealthRhythms' product, investigators will recruit 128 outpatients between the ages of 18 and 65, presenting to the University of Utah Department of Psychiatry outpatient clinics with a current mood and/or anxiety disorder. Sixty-four of these individuals will be randomly allocated to receive the full HealthRhythms package (Rhythm Sensing, Rhythm Trending, and Rhythm Stabilization) on their smartphones, while 64 will be asked to consent to Rhythm Sensing only. Participants in both arms will receive treatment as usual (TAU) for their mood and/or anxiety disorders, as typically provided at the University of Utah clinics. The duration of the study will be 16 weeks.

The primary outcome measures of the RCT will be the PROMIS Depression, the PROMIS Anxiety and the PROMIS Sleep Disturbance computerized adaptive testing (CAT) measures. The investigators hypothesize that those receiving the full package will demonstrate lower levels of depression, anxiety and sleep disturbance. In addition, investigators will explore the relationship between sensed rhythm stability and scores on patient-reported outcome measures of mood, anxiety and sleep disturbance (PROMIS). The investigators hypothesize that positive changes in the PROMIS measures will be mediated by positive changes in rhythm stability.

The primary outcome analyses will be based on random regression models, while the mediation analyses will follow the approach described by Helena Kraemer and colleagues.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-65
* Is currently in treatment for a mood and/or anxiety disorder, as defined by the DSM-5 (American Psychiatric Association, 2013).
* Patient participants need to be on a stable medication, however changes in dosage will be allowed during the course of this study
* Ability and willingness to give informed, written consent

Exclusion Criteria:

* Severe or poorly controlled concurrent medical disorders that may cause confounding depressive symptoms (e.g., untreated hypothyroidism or lupus) or require medication(s) that could cause depressive symptoms (e.g., high doses of beta blockers or alpha interferon)
* Meets criteria for one of the following concurrent DSM-5 psychiatric disorders: any organic or psychotic mental disorder other than bipolar disorder, current alcohol or drug dependence, primary obsessive compulsive disorder, primary eating disorder, or antisocial personality disorder
* Acute suicidal or homicidal ideation or requiring psychiatric hospitalization. Those who require inpatient treatment will be excluded (or discontinued) from the study and referred to for inpatient treatment.
* Cognitive deficits precluding use of a smartphone app and/or completion of patient-reported outcomes used at the University of Utah
* Insufficient fluency in English, provide clear verbal feedback about problems with the app, complete the study assessments, or make use of a smartphone app that involves very minimal instructions written in English.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 128 (Actual)
Dates: Start 2018-03-01 (Actual); Primary Completion 2019-05-31 (Actual); Study Completion 2020-07-31 (Actual)

PRIMARY OUTCOMES:
PROMIS Depression | Change at each timepoint (at 4, 8, 12, and 16 weeks)
  The PROMIS Depression instruments assess self-reported negative mood (sadness, guilt), views of self (selfcriticism, worthlessness), and social cognition (loneliness, interpersonal alienation), as well as decreased positive affect and engagement (loss of interest, meaning, and purpose)
PROMIS Anxiety | Change at each timepoint (at 4, 8, 12, and 16 weeks)
  The PROMIS Anxiety instruments measure self-reported fear (fearfulness, panic), anxious misery (worry, dread), hyperarousal (tension, nervousness, restlessness), and somatic symptoms related to arousal (racing heart, dizziness).
PROMIS Sleep | Change at each timepoint (at 4, 8, 12, and 16 weeks)
  The PROMIS Sleep Disturbance instruments assess self-reported perceptions of sleep quality, sleep depth, and restoration associated with sleep. This includes perceived difficulties and concerns with getting to sleep or staying asleep, as well as perceptions of the adequacy of and satisfaction with sleep

CONTACTS AND LOCATIONS:
Overall Officials: Ellen Frank, PhD, Principal Investigator — HealthRhythms, Inc.
Locations (1):
- University of Utah, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: Yes
The project will contain two distinct datasets: 1) data from HealthRhythms' collaboration with ImagineCare; and 2) data from the RCT of the Rhythm Stabilization Product (n=128). The investigators will not share the first dataset because it contains proprietary data not owned by HealthRhythms. The investigators will share the RCT data which will consist of self-reported measures, smartphone-sensed data and clinical assessments. Although the final dataset will be stripped of identifiers prior to sharing, there will remain a remote possibility of deductive disclosure of participants' identity using the sensed location data. The investigators will make the data and its documentation available to individuals via a data sharing agreement that requires a prior written commitment: 1) to only use the data for research purposes and not to identify participants; 2) to protect and secure the data using best practice security methods; and 3) to destroy the data once analysis has been completed.

REFERENCES:
- [Derived] Wallace ML, Frank E, McClung CA, Cote SE, Kendrick J, Payne S, Frost-Pineda K, Leach J, Matthews MJ, Choudhury T, Kupfer DJ. A translationally informed approach to vital signs for psychiatry: a preliminary proof of concept. NPP Digit Psychiatry Neurosci. 2024;2:14. doi: 10.1038/s44277-024-00015-8. Epub 2024 Aug 26. PMID 39639945
- [Derived] Frank E, Wallace ML, Matthews MJ, Kendrick J, Leach J, Moore T, Aranovich G, Choudhury T, Shah NR, Framroze Z, Posey G, Burgess SA, Kupfer DJ. Personalized digital intervention for depression based on social rhythm principles adds significantly to outpatient treatment. Front Digit Health. 2022 Sep 2;4:870522. doi: 10.3389/fdgth.2022.870522. eCollection 2022. PMID 36120713